CLINICAL TRIAL: NCT03145610
Title: Impact of a Triclosan-containing Toothpaste During the Progression of Experimental Peri-implant Mucositis: Clinical Parameters and Local Pattern of Osteo-immunoinflammatory Mediators in Peri-implant Fluid
Brief Title: Impact of a Triclosan-containing Toothpaste During the Progression of Experimental Peri-implant Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paulista University (Other)
Responsible Party: Principal Investigator, Fernanda Vieira Ribeiro, Professor, Paulista University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Triclosan Mucositis
Record Dates: First submitted 2017-04-27; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Biological Markers; Dental Implants; Cytokines; Triclosan; Toothpastes; Peri-Implantitis; Microbiology
MeSH Terms: conditions — Peri-Implantitis | interventions — Triclosan

STUDY DESIGN:
Intervention Model Description: This investigation was designed as double-blind, randomized, crossover study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo toothpaste (Placebo Comparator): Fluoride toothpaste will be used by filling the individual silicone stent allowing it to come into contact with the implant area for 2 min.
  Interventions: Other: Placebo toothpaste
- triclosan/copolymer/fluoride toothpaste (Experimental): triclosan/copolymer/fluoride toothpaste will be used by filling the individual silicone stent allowing it to come into contact with the implant area for 2 min.
  Interventions: Other: triclosan/copolymer/fluoride toothpaste

INTERVENTIONS:
Other: Placebo toothpaste — During an experimental 3-week period of undisturbed mechanical plaque accumulation in the implants, implants randomly assigned to Placebo group will be submitted to a chemical plaque control (three times per day) using a Triclosan toothpaste.
  Arms: Placebo toothpaste
Other: triclosan/copolymer/fluoride toothpaste — During an experimental 3-week period of undisturbed mechanical plaque accumulation in the implants, implants randomly assigned to triclosan/copolymer/fluoride group will be submitted to a chemical plaque control (three times per day) using a triclosan/copolymer/fluoride toothpaste.
  Arms: triclosan/copolymer/fluoride toothpaste

SUMMARY:
The aim of this study was to evaluate the influence of a triclosan-containing toothpaste in the profile of osteo-immunoinflammatory mediators in the peri-implant crevicular fluid (PICF) and in the clinical parameters during the progression of experimental peri-implant mucositis.

DETAILED DESCRIPTION:
Study design This investigation was designed as double-blind, randomized, crossover study to evaluate the influence of a triclosan-containing toothpaste in the profile of osteo-immunoinflammatory mediators in the PICF and in the clinical parameters during the progression of experimental peri-implant mucositis. This study was approved by the ethics committee of Paulista University (Protocol 97.117).

Population screening Patient recruitment started in June 2013 and was completed by the end of May 2014. The clinical procedures and evaluations were carried out between August 2013 and June 2014. Data entry and statistical analyses were performed in January 2015. All the patients in the study were recruited from the patients referred to Paulista University.

All eligible individuals were thoroughly informed of the nature, potential risks and benefits of their participation in the study, and they each signed an informed consent document.

Experimental groups During an experimental 3-week period of undisturbed plaque accumulation in the implants, patients were randomly assigned to two groups, according to chemical plaque control (three times per day): Triclosan (n=11): triclosan/copolymer/fluoride toothpaste or Placebo (n=11): fluoride toothpaste. Undisturbed plaque accumulation was achieved only in the nearby of dental implants by using an individual silicone tray involving the implant and adjacent teeth covering 2-3mm of peri-implant mucosa. The same silicone tray was filled by the respective toothpaste, according to the experimental group, during this period. Following 3 weeks, a professional prophylaxis was performed and a wash-out period of 30 days was established. Then, a second experimental 3-week period of undisturbed plaque accumulation in the implants was established and the experimental groups were exchanged. After that, a new professional prophylaxis was performed. All evaluations (clinical and immunoenzimatic assays) were performed at baseline, 3, 7, 14 and 21 days of each period of experimental mucositis induction.

The number of patients included in the present study was based on previous crossover investigations that found differences in the clinical parameters and crevicular fluid levels of osteo-immunoinflammatory markers in different clinical status.

Clinical examination The same examiner, who was blinded to the groups, performed all measurements of clinical assessment. To perform the intra-examiner calibration, 15 non-study individuals presenting dental implants were selected. The examiner measured the PD of all patients twice within 24 hours. The examiner was judged to be reproducible after fulfilling the pre-determined success criteria (the percentage of agreement within ± 1 mm between repeated measurements had to be at least 90%). The intra-class correlation was calculated as 92% reproducibility.

An individual stent was prepared to standardize the location of periodontal probe (North Carolina - Hu-Friedy, Chicago, IL, USA) to evaluate the following parameters at four sites of the experimental dental implants at baseline, 3, 7, 14, 21 days follow-ups: 1) plaque index (PI/%): scored using a dichotomous plaque index along the mucosal margin around implants, 2) bleeding index (BI/%): scored using dichotomous index of mucosal marginal bleeding around implants, 3) Position of the peri-implant margin (PPM/mm), which was the distance from the stent to the peri-implant margin; 4) Relative clinical attachment level (RCAL/mm), which was the distance from the stent to the bottom of the peri-implant pocket; and 5) Peri-implant probing depth (PD/mm), calculated by deducting PPM from RCAL. The full mouth plaque scores (FMPS) and bleeding scores (FMBS) were calculated before the beginning of each period of experimental mucositis induction.

Osteo-immunoinflammatory profile assessment Peri-implant crevicular fluid was collected from dental implant sites by the same examiner. The area was isolated, dried and fluid was collected at two sites of the experimental dental implants (vestibular and lingual) by placing filter paper strips (Periopaper, Oraflow, Plainview, NY, USA) into the sulcus until the clinician perceived a slight resistance, and then leaving in place for 15 s. The fluid volume was measured with a calibrated device (Periotron 8000, Oraflow, Plainview, NY, USA). The strips were placed into sterile tubes containing 400 μL of phosphate-buffered saline (PBS) with 0.05% Tween-20. Peri-implant crevicular fluid samples were immediately stored at -20 °C.

Levels of interferon (INF), interleukin (IL)-4, IL-17, IL-1β, IL-10, IL-6, IL-23, tumor necrosis factor (TNF)-α (Human Th17 HTH17MAG-14K, Millipore Corporation, Billerica, MA, USA), osteoprotegerin (OPG), osteocalcin (OC), osteopontin (OPN) (Human Bone HBNMAG-51K, Millipore Corporation, Billerica, MA, USA), matrix metalloproteinase (MMP)-2, MMP-9 (Human MMP Panel 2 HMMP2MAG-55K, Millipore Corporation, Billerica, MA, USA), transforming growth factor (TGF)-β (Multi-species TGFβ TGFBMAG-64K, Millipore Corporation, Billerica, MA, USA) and crosslinked telopeptide of type I collagen (ICTP) (Uscn Life Science Inc. Wuhan, Hubei, PRC) in the peri-implant fluid were determined using commercially available kits. Assays were carried out according to the manufacturer's recommendations using the MAGpix™ instrument (MiraiBio, Alameda, CA, USA). The samples were individually analyzed, and concentrations were estimated from the standard curve using a five-parameter polynomial equation using Xponent® software (Millipore, Corporation, Billerica, MA, USA). The mean concentration of each mediator was calculated using the individual as a statistical unit and expressed as pg/ml.

Data analysis All analyses were performed using SAS program release 9.1 (Cary, NC, USA). Data were firstly examined for normality using the Kolmogorov-Smirnov test, and the data that achieved normality were analysed using parametric methods. The percentages of experimental sites with visible plaque accumulation, BI and the PD means were computed for each implant selected for peri-implant fluid sampling. Subsequently, clinical parameters and the local levels of osteo-immunoinflammatory mediators were averaged into Placebo and Triclosan groups. The differences in FMPS and FMBS - measured before the beginning of each period of experimental mucositis induction.- between both groups were compared using the Wilcoxon test. For the other clinical parameters (PI, BI, PPM, RCAL and PD), ANOVA/Tukey test was used to detect differences between groups and periods. Concentrations of osteo-immunoinflammatory markers between groups and among follow-ups were compared using the Wilcoxon and Friedman test, respectively. An experimental level of significance was determined at 5% for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* 30 years old or more
* present at least a 2-stage unitary screwed implant-supported single-unit crown in the molar or pre-molar region
* implant connection should be external hexagonal and the implants should be in function at least 12 months with width of keratinized tissue > 2mm around implants
* The peri-implant tissue should be healthy [probing depth (PD) <4mm with no bleeding on probing (BoP) and no evidence of radiographic bone loss beyond bone remodeling (AAP 2013).
* Patients should be periodontally healthy and present full mouth plaque scores (FMPS, Ainamo & Bay 1975) and bleeding score (FMBS, Muhlemann & Son 1971) < 20%.

Exclusion Criteria:

* pregnancy
* lactation
* smokers
* systemic conditions r that could affect the progression of peri-implant diseases and bone metabolism (e.g., immunologic disorders), use of long-term administration of anti-inflammatory and immunosuppressive medications
* antibiotic therapies in the previous 6 months
* individuals that required bone grafts before or alongside the implant surgery
* history of previous regenerative procedures in the area treated with implant therapy.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2014-05-30 (Actual); Study Completion 2015-01-14 (Actual)

PRIMARY OUTCOMES:
bleeding index | 21 days
  scored using dichotomous index of mucosal marginal bleeding around implants,

SECONDARY OUTCOMES:
plaque index | 21 days
  scored using a dichotomous plaque index along the mucosal margin around implants
Position of the peri-implant margin | 21 days
  distance from the stent to the bottom of the peri-implant pocket;
Peri-implant probing depth | 21 days
  calculated by deducting PPM from RCAL
Relative clinical attachment level | 21 days
  which was the distance from the stent to the bottom of the peri-implant pocket;
Osteo-immunoinflammatory mediators | 21 days
  Levels of interferon (INF), interleukin (IL)-4, IL-17, IL-1β, IL-10, IL-6, IL-23, tumor necrosis factor (TNF)-α (Human Th17 HTH17MAG-14K, Millipore Corporation, Billerica, MA, USA), osteoprotegerin (OPG), osteocalcin (OC), osteopontin (OPN) (Human Bone HBNMAG-51K, Millipore Corporation, Billerica, MA, USA), matrix metalloproteinase (MMP)-2, MMP-9 (Human MMP Panel 2 HMMP2MAG-55K, Millipore Corporation, Billerica, MA, USA), transforming growth factor (TGF)-β (Multi-species TGFβ TGFBMAG-64K, Millipore Corporation, Billerica, MA, USA) and crosslinked telopeptide of type I collagen (ICTP) (Uscn Life Science Inc. Wuhan, Hubei, PRC) in the peri-implant fluid were determined using commercially available kits.

IPD SHARING:
Plan to Share IPD: No